CLINICAL TRIAL: NCT06583096
Title: College Student Stress: Transitions Over Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Adam Horwitz, Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00257547; K23MH131761 (NIH)
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Depressive Symptoms
Keywords: First-year college student; Surveys; Supportive text messages; Stress; Personalized feedback
MeSH Terms: conditions — Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: After initial survey (screening) is received, participants that are eligible for the trial and complete the baseline assessments will be assigned (3:1) to the "Assessment Only" (n = 30) or the "Intervention" (n=90) condition".
  The intervention arm contains two components: personalized feedback reports and supportive text messages. Each week participants are randomized, with a 2:1 probability to receive (versus not receive) a personalized feedback report, and a 2:1 probability to receive (versus not receive) supportive text messages during the week. For those randomized to receive text messages in a given week, there is a daily 50:50 randomization to receive (or not receive) a text message.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment Only (Other): Weekly surveys only.
  Interventions: Behavioral: Surveys
- Intervention - surveys, text messages, and feedback reports (Experimental): Participants in the intervention arm will be randomized to receive (or not receive) text messages in a given week, with a daily randomization to receive (or not receive) a text message if randomized to receive text messages that week.
  Additionally, participants will be randomized each week to receive (or not receive) personalized feedback reports.
  Interventions: Behavioral: Surveys; Behavioral: Supportive Text messages; Behavioral: Personalized Feedback (PF) Report

INTERVENTIONS:
Behavioral: Surveys — Participants (in both arms) will complete surveys once per week and participants in the intervention arm will also complete additional 1-minute surveys daily. Study participation will be completed at the conclusion of the final follow-up survey administered 6-weeks after study enrollment.
Behavioral: Supportive Text messages — Text messages will be sent Mondays-Sunday if participants are randomized to receive them in a given week, with a daily 50:50 send/no-send randomization. A bank of 25 text messages will be used for the study, providing tips/strategies across a range of topics, including managing time and academic stressors, recommendations for self-care and mood management, and messages geared towards fostering social connections and support. Some messages will contain links to videos, websites, or articles for more information on a topic.
  Arms: Intervention - surveys, text messages, and feedback reports
Behavioral: Personalized Feedback (PF) Report — For individuals that are randomized to receive a Personalized Feedback Report, the study team will send participants a text on a Monday with the feedback from the prior survey (baseline survey in the first week, weekly survey in the next five weeks). There will be graphs for depression, anxiety, stress, and flourishing.
  Arms: Intervention - surveys, text messages, and feedback reports

SUMMARY:
This research study is being conducted to better understand how college students develop and cope with stress and to identify opportunities to help students notice and respond to stress early before symptoms contribute to significant negative consequences.

This project will be completed in two parts. In the first part (not a trial) participants will be asked to complete a screening survey to determine eligibility. Eligible participants (i.e., those with mild-to-moderate depressive symptoms and not receiving mental health care) will continue into the clinical trial portion (part two). There were 120 students in the clinical trial phase of the study, where 30 were randomly assigned to "assessment only" and 90 to the "intervention" condition.

ELIGIBILITY:
Inclusion Criteria:

* First-year college students that are full-time or part-time students enrolled at the University of Michigan, Ann Arbor or Flint campuses
* Mild-to-moderate depressive symptoms, and are not receiving professional mental health services will be eligible

Exclusion Criteria:

* Under the age of 17
* Currently be receiving mental health therapy/counseling from a healthcare professional
* Experiencing minimal depressive symptoms (defined in protocol)
* Experiencing moderately severe to severe depressive symptoms (defined in protocol)

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Horwitz, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared upon request following publication of primary results.
Supporting Information: Study Protocol, ICF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 353 individuals were consented to be screened for participant eligibility, and 126 were determined to be eligible for the randomized trial portion.
Pre-assignment Details: Of the 126 individuals eligible to be randomized, 120 agreed to become randomized participants.
Groups:
- Assessment Only: Participants completed assessment surveys once per week over six weeks.
- Intervention: Participants completed assessment surveys once per week over six weeks. Participants in this arm also completed brief (1-minute) daily surveys during this period. Participants in the intervention arm were randomized to receive (or not receive) text messages in a given week, with a daily randomization to receive (or not receive) a text message if randomized to receive text messages that week. Additionally, participants were randomized each week to receive (or not receive) personalized feedback reports.
Period: Overall Study
Arm/Group | Assessment Only | Intervention
Started | 30 | 90
Completed (Participants were completers if they completed the 6-week follow-up assessment.) | 26 | 78
Not Completed | 4 | 12
Not completed — Lost to Follow-up | 4 | 10
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Only eligible individuals who were randomized had baseline data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Assessment Only | Intervention | Total
Number analyzed (Participants) | 30 | 90 | 120
Age, Customized [Count of Participants; unit: Participants]
  17 years | 4 | 12 | 16
  18 years | 23 | 67 | 90
  19 years | 3 | 9 | 12
  20 - 25 years | 0 | 2 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 10 | 28 | 38
  Female | 19 | 58 | 77
  Transgender/Non-binary | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 27 | 81 | 108
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 17 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 7 | 9
  White | 23 | 53 | 76
  More than one race | 2 | 11 | 13
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 90 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Participants Who Agreed to Participate in the Trial
Description: Of the individuals meeting eligibility criteria (i.e., mild-to-moderate depressive symptoms, no current mental health service utilization) from the initial screen, what percentage agreed to be enrolled and randomized into the clinical trial.
Time Frame: Up to 10 days after screening survey
Population: Analysis of this outcome measure occurred prior to randomization. 126 participants were eligible prior to randomization.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: Participants completed the screen and were eligible for enrollment and subsequent randomization
Arm/Group | Eligible Participants
Number analyzed (Participants) | 126
Participants | 120

2. Primary Outcome: Percentage of Participants Who Completed Follow-ups
Description: Weekly ten-minute surveys assessing mental health symptoms, stress, and adaptive functioning were sent to participants. Results reflect the number of participants who completed their survey each week.
Time Frame: Baseline up to six-week follow-up
Population: Some participants did not complete weekly surveys consecutively.
Measure: Count of Participants; unit: Participants
Arm/Group | Assessment Only | Intervention
Number analyzed (Participants) | 30 | 90
Participants
  Week 1 | 23 | 81
  Week 2 | 23 | 80
  Week 3 | 24 | 79
  Week 4 | 25 | 78
  Week 5 | 24 | 76
  Week 6 | 26 | 78

3. Primary Outcome: Percentage of Participants That Remain Active (i.e. do Not Request to Stop Messages) on the Text-message Group
Description: Results reflect the participants who remained active during the full trial in the intervention group.
Time Frame: Baseline up to six-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 90
Participants | 88

4. Primary Outcome: Number of Withdrawals
Description: Results reflect participants who requested to withdraw from the trial.
Time Frame: Baseline up to six-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Assessment Only | Intervention
Number analyzed (Participants) | 30 | 90
Participants | 0 | 2

5. Primary Outcome: Total Percent of Feedback Reports That Were Viewed Across All Sent Feedback Reports
Description: As part of the intervention arm, participants were randomized each week to receive or not receive personalized feedback reports. Reports had graphical explanations of the participant's responses to the survey questions. The data values reported reflect the number of participants who viewed feedback reports, while the Number Analyzed for each Row reflects the number of participants who were sent a personalized feedback report that week.
Time Frame: Baseline up to six-week follow-up
Population: Not all participants were sent the feedback reports each week.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Surveys, Text Messages, and Feedback Reports
Number analyzed (Participants) | 90
Participants
  Week 1: number analyzed (Participants) | 60
  Week 1 | 37
  Week 2: number analyzed (Participants) | 61
  Week 2 | 34
  Week 3: number analyzed (Participants) | 62
  Week 3 | 29
  Week 4: number analyzed (Participants) | 66
  Week 4 | 30
  Week 5: number analyzed (Participants) | 54
  Week 5 | 26
  Week 6: number analyzed (Participants) | 60
  Week 6 | 29

6. Primary Outcome: Percent of Participants (in the Intervention Arm) That Viewed a Personalized Feedback Report at Least Once
Description: As part of the intervention, some participants in the intervention arm were randomly sent feedback reports. Reports had graphical explanations of the participant's response to the survey questions. All participants in the intervention arm were sent at least one feedback report during the course of the trial. Results reflect the number of participants who viewed at least one report.
Time Frame: Baseline up to six-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Surveys, Text Messages, and Feedback Reports
Number analyzed (Participants) | 90
Participants | 70

7. Primary Outcome: Participant Self-reported Satisfaction With the Intervention Components - Assessment-only
Description: Participants in the "Assessment Only" arm who completed the 6-week follow-up survey responded to an 8-question survey regarding their satisfaction with the study. Each question was on a scale of 1 to 7 (1-Strongly disagree, 4 Neither agree nor disagree, 7-Strongly Agree). A higher score indicated more satisfaction with the study. Results reflect the average participant scores for each question.
Time Frame: Six-week follow-up
Population: This includes the 26 (of 30) participants who completed the 6-week follow-up survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assessment Only
Number analyzed (Participants) | 26
units on a scale
  I am glad I participated in the study. | 6.12 (0.77)
  The weekly Sunday surveys helped me to reflect on how things were going in my life. | 6.00 (0.82)
  I would be willing to complete brief (~5 minute) weekly surveys during the year without compensation | 3.24 (1.64)
  My confidentiality and privacy was respected during this study. | 6.20 (0.87)
  Six weeks was too brief for this study period. | 4.12 (1.30)
  Participating in this study was beneficial for my health and well-being. | 5.16 (1.14)
  The system of receiving messages and completing surveys was convenient. | 6.40 (0.91)
  I liked participating in this study. | 6.04 (1.02)

8. Primary Outcome: Participant Self-reported Satisfaction With the Intervention Components - Intervention Only
Description: Participants in the "Intervention" arm who completed the 6-week follow-up survey responded to an 18-question survey regarding their satisfaction with the intervention. Each question was on a scale of 1 to 7 (1-Strongly disagree, 4 Neither agree nor disagree, 7-Strongly Agree). A higher score indicated more satisfaction. Results reflect the average participant scores for each question.
Time Frame: Six-week follow-up
Population: This included the 78 (of 90) participants who completed the 6-week follow-up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 78
score on a scale
  I am glad that I participated in this study. | 6.18 (1.00)
  The daily 5-item surveys helped me to reflect on how things were going in my life. | 5.90 (1.11)
  The coping/support text-message strategies were useful for me. | 4.31 (1.73)
  I would be willing to complete brief (~5 minute) weekly surveys during the year without compensation | 4.04 (1.71)
  The personalized feedback reports provided valuable insight into how I was doing over time. | 5.25 (1.23)
  The number of coping/support text messages I received was… (1-too few, 4-just right, 7-too many) | 4.18 (1.36)
  Six weeks was too brief for this study period. | 4.26 (1.41)
  Participating in this study was beneficial for my health and well-being. | 5.18 (0.93)
  I would have liked to receive personalized feedback graphs every week. | 4.75 (1.48)
  The weekly Sunday surveys helped me to reflect on how things were going in my life. | 5.51 (0.94)
  I would be willing to complete brief (~1 minute) daily surveys during the year without compensation. | 4.03 (1.62)
  The study's intervention meets my approval. | 5.35 (0.98)
  The system of receiving messages and completing surveys was convenient. | 6.09 (0.81)
  The study's intervention was appealing to me. | 5.44 (0.99)
  A program like this study should be offered to all students. | 5.61 (1.16)
  I would want to continue receiving surveys, texts, and personalized feedback reports after the study | 4.12 (1.58)
  I like the intervention from this study. | 5.12 (1.00)
  My confidentiality and privacy was respected during this study. | 5.97 (0.90)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Assessment Only | Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/90
Other Adverse Events (participants affected / at risk) | 7/30 | 17/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Assessment Only (N=30) | Intervention (N=90)
Moderately severe to severe depression (Psychiatric disorders) | 7 | 13
Suicidal ideation in the past week (Psychiatric disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT06583096/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT06583096/ICF_000.pdf